CLINICAL TRIAL: NCT02527863
Title: The Effects of Tolvaptan on Renal Handling of Water and Sodium, Vasoactive Hormones and Central Hemodynamics During Baseline Conditions and After Inhibition of the Nitric Oxide System in Patients With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Effect of the Aquaretic Tolvaptan on Nitric Oxide System
Acronym: TOPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, Professor, MD, Dr.Sci., Regional Hospital Holstebro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SAFA-2-2014; 2014-001973-15 (EudraCT Number)
Record Dates: First submitted 2015-02-18; First posted 2015-08-19 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Tolvaptan; L-NMMA; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 60 mg Tolvaptan (Active Comparator): Oral administration of 60 mg tolvaptan on each examination day.
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator): Oral administration of a Unikalk tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan — 60 mg Tolvaptan pr day for 1 day
  Other Names: Samsca
  Arms: 60 mg Tolvaptan
Drug: Placebo — 1 tablet Unikalk pr day for 1 day
  Other Names: Unikalk
  Arms: Placebo

SUMMARY:
Tolvaptan is a selective vasopressin receptor antagonist (V2R) that increases free water and sodium excretion. Inhibition of V2R increases vasopressin concentration in plasma, which stimulates V1-receptors in the vascular bed and may change both central and brachial hemodynamics and plasma concentration of vasoactive hormones.

The purpose of the study is to measure the effects of tolvaptan on renal handling of water and sodium, systemic hemodynamics and vasoactive hormones at baseline and during nitric oxide (NO)-inhibition with L-NG-monomethyl-arginine (L-NMMA) in patients with autosomal dominant polycystic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian men and women
2. Age between 18-65 years
3. ADPKD, diagnosed by genetic testing of PKD1 (>85%) or PKD2 mutations, or by ultrasonography:

   1. patients with negative family history for ADKPD and more than 10 cysts in each kidney and no extrarenal or renal findings that suggest causes to cyst formation.
   2. patients with positive family history for ADPKD:

      * 15-39 yr of age and at least 3 or more unilateral or bilateral.
      * 40-59 yr of age and 2 or more cysts in each kidney.
      * 60 yr of age and at least 4 cysts in each kidney.
4. Kidney function corresponding to CKD stages 1-3(eGFR> 30 mL/min/1,73 m2),
5. BMI between 18.5 and 35.5 kg/m2.

Exclusion Criteria:

1. Clinical signs of diseases in the heart, lungs, endocrine organs, brain or neoplastic disease,
2. clinically significant abnormalities in blood or urine sample at the inclusion
3. previous cerebrovascular insults,
4. previous clinical evidence for aneurysm
5. Alcohol or drug abuse,
6. smoking,
7. pregnancy or breastfeeding,
8. clinically significant changes in the electrocardiogram,
9. medication except antihypertensive agents and oral contraceptives,
10. blood pressure>170/105 mmHg despite treatment with metoprolol and/or amlodipine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
CH2O (Measurement of H2O clearance) | 5-6 Hours
  Measurement of H2O clearance at baseline, during and after L-NMMA infusion

SECONDARY OUTCOMES:
Urine biomarkers(Aquaporins and Epithelial Sodium Channels γ) | 5-6 Hours
Central and brachial blood pressure | 5-6 Hours
Augmentation Index | 5-6 Hours
Vasoactive Hormones( Angiotensin II, Aldosterone, Endothelin, Atrial Natriuretic Peptide, Brain Natriuretic Peptide, Arginin Vasopressin) | 5-6 Hours
Fractional sodium excretion | 5-6 Hours
  Measurement of Sodium excretion at baseline, during and after L-NMMA infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Study Chair — Department of Medical Research and Medicine, Holstebro Regional Hospital Holstebro, Holstebro, Denmark, 7500
Locations (1):
- Department of Medical Research and Medicine, Holstebro Regional Hospital, Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Al Therwani S, Malmberg MES, Rosenbaek JB, Bech JN, Pedersen EB. Effect of tolvaptan on renal handling of water and sodium, GFR and central hemodynamics in autosomal dominant polycystic kidney disease during inhibition of the nitric oxide system: a randomized, placebo-controlled, double blind, crossover study. BMC Nephrol. 2017 Aug 15;18(1):268. doi: 10.1186/s12882-017-0686-3. PMID 28810844